CLINICAL TRIAL: NCT05570110
Title: Double-blind Randomized Placebo Controlled Study on the Effect of Enoxolone ( 11-beta Hydroxysteroid-dehydrogenase Type 2 Inhibitor) on the RAAS, Autonomic and Imaging Biomarkers and the Outcome of Depression
Brief Title: Enoxolone in Major Depression - Biomarker-outcome Relationship
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: Slovak Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Harald Murck, Apl. Professor, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MNS_02.1
Record Dates: First submitted 2022-09-28; First posted 2022-10-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Unipolar Depression
Keywords: Atypical depression;
MeSH Terms: conditions — Depressive Disorder | interventions — Glycyrrhetinic Acid

STUDY DESIGN:
Intervention Model Description: Randomized parallel group design, first two subjects open label.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active and Placebo Capsules of the same shape and size are utilized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- enoxolone (Experimental): 100 mg enoxolone in a capsule
  Interventions: Drug: Enoxolone
- placebo (Placebo Comparator): Placebo in a capsule
  Interventions: Drug: Enoxolone

INTERVENTIONS:
Drug: Enoxolone — one capsule of active or placebo in the evening
  Other Names: glycyrrhetinic acid

SUMMARY:
Many different forms of depression exist. It is difficult to predict to what treatment a given patient with depression responds. Studies demonstrate that biomarkers can help to distinguish different forms of depression. Simple markers, like aldosterone/cortisol in body fluids, blood pressure and inflammation markers , have been identified as predictors of therapy resistance in depression. Enoxolone is a molecule derived from the licorice plant and has demonstrated an effect on these biomarkers, which may imply an improved response. The current randomized placebo controlled study is assessing whether the presence of markers of therapy resistance can predict a preferential effect of enoxolone vs. placebo on clinical outcome. Secondarily, it is tested whether these markers change differentially in the treatment groups. Finally, the relationship between the change of the markers and clinical change will be assessed.

DETAILED DESCRIPTION:
The objective of the study is 1. to confirm patient characteristics, which are related to lesser responsivity to antidepressant treatment and 2. to explore the utility of the 11-beta hydroxysteroid-dehydrogenase type 2 (11betaHSD2) and toll-like receptor (TLR)-4 inhibitor enoxolone to reverse these markers of refractoriness and, potentially, improve clinical outcome. A broad spectrum of patients is recruited in order to provide the opportunity to compare those with relevant markers of refractoriness vs. those without.

The identified markers are related to the activity of aldosterone, which appears to affect specific CNS areas, which are involved in mood and autonomic regulation. One area of particular relevance is the pontine nucleus of the solitary tract (NTS). Potential primary triggers for an increased aldosterone release under stressful conditions are related to low blood pressure, electrolyte alterations and a dysfunction of the peripheral mineralocorticoid receptor (MR). The resultant aldosterone release evokes activity at the NTS, which may lead to depression and anxiety.

Enoxolone leads to an activation primarily of the peripheral MR by reducing the activity of the 11betaHSD2, therefore allowing cortisol access to the MR and, as a consequence, suppress the release of renin, angiotensin and aldosterone. In addition, it can increase blood pressure slightly.

1. A set of potentially predictive markers for therapy response of enoxolone vs. placebo will be studied, based on this mechanistic pathway, in detail:

   For the primary analysis subjects are grouped into those with higher vs. lower systolic blood pressure values, as determined by the median systolic blood pressure value at baseline.

   For the secondary analysis the ratio of urine aldosterone/cortisol, as collected over night will be used as a differentiating parameter. Split at the median defines the groups.

   Exploratory parameters for a split are the following:
   1. sleep duration
   2. heart rate variability
   3. salt taste sensitivity and salt preference
   4. inflammation markers, in particular C-reactive protein in plasma.
   5. Optional: volumes of lateral ventricles, corpus callosum and choroid plexi.
   6. Optional: white matter integrity, as measured by diffusion tensor imaging
2. Markers of target engagement:

   1. Effect of enoxolone vs. placebo on systolic blood pressure.
   2. Effect of enoxolone vs. placebo on urine aldosterone/cortisol concentration.
   3. Effect of enoxolone vs. placebo on plasma sodium/potassium concentration ratio.
   4. Effect of enoxolone on C-reactive protein and other inflammation markers.
3. The relationship between changes in hormone concentrations and markers of CNS activation of MR, i.e. functional CNS target engagement. These are:

   1. Heart rate variability and heart rate
   2. Systolic blood pressure at rest and nocturnal blood pressure dip
   3. Total sleep time
   4. Salt taste preference and sensitivity
   5. Inflammatory markers
   6. Optional: volumes of lateral ventricles, corpus callosum and choroid plexi.
   7. Optional: white matter integrity, as measured by diffusion tensor imaging

ELIGIBILITY:
Inclusion Criteria:

* Unipolar Depression
* in women: Contraceptive means

Exclusion Criteria:

* Schizophrenic and delusional disorders
* Neurological diseases in which central nervous system involvement is known, such as epilepsies, storage diseases; severe mental retardation
* Internistic diseases of moderate or higher severity, which may make participation in the study risky from a clinical point of view. In particular, multiple systolic blood pressure (measured after at least 5 min supine position) of > 145 mm Hg as well as hypokalemia (< 3.5 mmol/l) and clinically relevant ECG changes
* Poorly controlled diabetes mellitus (HbA1c > 10)
* Pregnancy or active desire for pregnancy for the duration of the study
* Non-consent or inability to consent to the study
* Treatment with the following substances: spironolactone or eplerenone; systemic glucocorticoids
* Treatment with ketamine or electroconvulsive therapy in the last 3 months before randomization
* Acute suicidality
* Intolerance to licorice preparations or licorice contents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Plasma and urine aldosterone/cortisol ratio | Baseline, as predictor for differentiation of treatment groups clinical response
  ratio of plasma aldosterone/cortisol at awakening; ratio of nocturnal urine aldosterone concentration/urine cortisol concentration
C-reactive protein | Baseline, as predictor for differentiation of treatment groups clinical response and change from baseline (4 weeks)
  C-reactive protein in plasma
Systolic blood pressure | Baseline, as predictor for differentiation of treatment groups clinical response
  Systolic blood pressure at rest at baseline as a predictor for treatment differentiation
Depression rating | change from baseline to week 4, with systolic blood pressure as covariate
  Hamilton depression rating scale (HAMD) - 17 items; higher is worse

SECONDARY OUTCOMES:
Urine aldosterone/cortisol ratio | change from baseline to week 4
  Ratio of nocturnal urine aldosterone concentration/urine cortisol concentration
Plasma ratio of sodium/potassium | change from baseline to week 4
  Ratio of the plasma concentration of sodium/ plasma concentration of potassium
Nocturnal heart rate variability | change from baseline to week 4
  Average nocturnal heart rate variability, expressed as stress level (Garmin, arbitrary unit)
Nocturnal blood pressure dip (difference between pre-sleep and minimal nocturnal blood pressure | change from baseline to week 4
  Minimum of continuously monitored systolic blood pressure (mmHg)
Depression self rating | change from baseline to week 4
  Patient health questionnaire-9 (PHQ-9), higher is worse
Total sleep duration | change from baseline to week 4
  Total sleep duration, as determined by wearable device (Garmin) (minutes)
Salt taste preference and sensitivity | change from baseline to week 4
  salt taste preference, as determined by tasting a 0.9% NaCl solution, 11 item Likert scale (Murck et al., 2018)
Rating for symptoms of normal pressure hydrocephalus | change from baseline to week 4
  Idiopathic normal pressure hydrocephalus grading scale (iNPHGS) (Kubo et al., 2008), higher is worse

OTHER OUTCOMES:
Lateral cerebral ventricular volume | change from baseline to 4 weeks
  Volume of lateral ventricles (sum) (mL), measured by MRI with freesurfer program
Corpus callosum volume | change from baseline to 4 weeks
  Volume of corpus callosum (mL) segments, measured by MRI with freesurfer program
Choroid Plexus Volume | change from baseline to 4 weeks
  Volume of Choroid Plexi (sum) (mL), measured by MRI with freesurfer program
Saliva cortisol ratio | change from baseline to 4 weeks
  Ratio of saliva cortisol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Harald Murck, MD PhD, Study Director — Philipps University Marburg
Locations (1):
- Clinic for Psychiatry and Psychotherapy, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Plan to share study data in concordance with local regulations
Supporting Information: Study Protocol
Time Frame: available after study completion
Access Criteria: CDA or other agreements

REFERENCES:
- [Background] Murck H. Discovery of Personalized Treatment for Immuno-Metabolic Depression-Focus on 11beta Hydroxysteroid Dehydrogenase Type 2 (11betaHSD2) and Toll-like Receptor 4 (TLR4) Inhibition with Enoxolone. Pharmaceuticals (Basel). 2025 Oct 10;18(10):1517. doi: 10.3390/ph18101517. PMID 41155634
- [Background] Murck H, Luerweg B, Hahn J, Braunisch M, Jezova D, Zavorotnyy M, Konrad C, Jansen A, Kircher T. Ventricular volume, white matter alterations and outcome of major depression and their relationship to endocrine parameters - A pilot study. World J Biol Psychiatry. 2021 Feb;22(2):104-118. doi: 10.1080/15622975.2020.1757754. Epub 2020 May 15. PMID 32306867
- [Background] Murck H, Lehr L, Hahn J, Braunisch MC, Jezova D, Zavorotnyy M. Adjunct Therapy With Glycyrrhiza Glabra Rapidly Improves Outcome in Depression-A Pilot Study to Support 11-Beta-Hydroxysteroid Dehydrogenase Type 2 Inhibition as a New Target. Front Psychiatry. 2020 Dec 10;11:605949. doi: 10.3389/fpsyt.2020.605949. eCollection 2020. PMID 33362613
- [Background] Engelmann J, Murck H, Wagner S, Zillich L, Streit F, Herzog DP, Braus DF, Tadic A, Lieb K, Muller MB. Routinely accessible parameters of mineralocorticoid receptor function, depression subtypes and response prediction: a post-hoc analysis from the early medication change trial in major depressive disorder. World J Biol Psychiatry. 2022 Oct;23(8):631-642. doi: 10.1080/15622975.2021.2020334. Epub 2022 Jan 25. PMID 34985381
- [Background] Murck H, Braunisch MC, Konrad C, Jezova D, Kircher T. Markers of mineralocorticoid receptor function: changes over time and relationship to response in patients with major depression. Int Clin Psychopharmacol. 2019 Jan;34(1):18-26. doi: 10.1097/YIC.0000000000000239. PMID 30300165